CLINICAL TRIAL: NCT01508689
Title: Effect of Calcium-fortified Cereal Bars on Dietary Calcium Intake in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 16802
Record Dates: First submitted 2012-01-09; First posted 2012-01-12 (Estimated); Last update posted 2015-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Calcium Deficiency
Keywords: Cereal bar; Calcium-fortified; Calcium intake

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Receive cereal bars first (Other): This group will receive Kellogg's Nutri-Grain® cereal bars during the second three weeks of the study.
  Interventions: Behavioral: Receive Kellogg's Nutri-Grain® cereal bars first
- Receive cereal bars second (Other): This group will receive Kellogg's Nutri-Grain® cereal bars during the last three weeks of the study.
  Interventions: Behavioral: Receive Kellogg's Nutri-Grain® cereal bars second

INTERVENTIONS:
Behavioral: Receive Kellogg's Nutri-Grain® cereal bars first — First three weeks of study: consume perceived usual diet; Second three weeks of study: Receive 42 Kellogg's Nutri-Grain® cereal bars per person, consume 2 bars per day; Third three weeks of study: consume perceived usual diet
  Arms: Receive cereal bars first
Behavioral: Receive Kellogg's Nutri-Grain® cereal bars second — First six weeks of study: consume perceived usual diet; Last three weeks of study: Receive 42 Kellogg's Nutri-Grain® cereal bars per person, consume 2 bars per day
  Arms: Receive cereal bars second

SUMMARY:
The purpose of this study is to determine whether eating Kellogg's Nutri-Grain cereal bars will increase calcium intake in healthy adult women.

DETAILED DESCRIPTION:
The average intake of calcium in women in the United States from the diet (about 800 mg/day) is below the Recommended Dietary Allowance (1000 mg/day for ages 18 to 50 years, 1200 mg/day for age above 50 years), which increases their risk of developing osteoporosis. Consumption of two calcium-fortified cereal bars per day may be a feasible way to increase the dietary intake of calcium. This study will use Kellogg's Nutri-Grain® cereal bars, which provide 200 mg of calcium per bar, or a total of 400 mg/day.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Able to speak, read, and understand English
* Able to consume Kellogg's Nutri-Grain® cereal bars

Exclusion Criteria:

* Consumption of calcium supplements or calcium-containing medications
* Regular consumption of 2 Kellogg's Nutri-Grain® cereal bars per month
* Currently pregnant or planning to become pregnant during the course of the study
* Liver disease
* Kidney disease
* Gastrointestinal disease (celiac disease, ulcerative colitis, or Crohn's disease)
* Have a history of bariatric surgery
* Had a major cardiovascular event (stroke or myocardial infarction)
* Undergoing treatment of cancer with the exception of non-melanoma cancer
* Following a weight control diet, a disease specific diet, or a vegan diet
* Have a diagnosed eating disorder
* Allergic to any of the ingredients in the study bar

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2012-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Dietary calcium intake | 9 weeks
  1 form of 3-day diet diary per week will be assessed during weeks 2, 6, and 8 of study

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Lee, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Houston, Texas, United States

REFERENCES:
- [Derived] Lee JT, Moore CE, Radcliffe JD. Consumption of calcium-fortified cereal bars to improve dietary calcium intake of healthy women: randomized controlled feasibility study. PLoS One. 2015 May 5;10(5):e0125207. doi: 10.1371/journal.pone.0125207. eCollection 2015. PMID 25941810